CLINICAL TRIAL: NCT06884137
Title: Investigation of the Relationship Between Neck Pain and Spinal Curvatures in Patients With Chronic Neck Pain
Brief Title: Investigation of the Relationship Between Neck Pain and Spinal Curvatures
Acronym: neck pain
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Buket Büyükturan, Kırşehir Ahi Evran Univercity, Kirsehir Ahi Evran Universitesi
Other Study IDs: 28.06.2012/4271/223
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain
Keywords: spinal curvatures; neck pain
MeSH Terms: conditions — Neck Pain; Spinal Curvatures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the Experimental group: Individuals with neck pain score of 5 or less according to Visual Analogue Scale (VAS) were identified as Group 1
- the control group: Individuals with neck pain score of 5 or less according to Visual Analogue Scale (VAS) were identified as Group 1, whereas those with any score above 5 were identified as Group 2.

SUMMARY:
Although it is known that the cervical, thoracic and lumbar regions of the spine are related with each other biomechanically, there are no studies examining the relationship between cervical pain and other regions of the spine. The purpose of this study was to examine angular changes of the spine and compare it with the control group according to the state of pain in patients with neck pain.

81 patients with chronic neck pain and 40 without any pain in their neck were included in the study. Spinal Mouse device was used to evaluate thoracic and lumbar curvatures. The pain sensory was evaluated with VAS.

DETAILED DESCRIPTION:
Neck pain is one of the most common problems among musculoskeletal disorders. Individuals with recurrent neck pain are characterized with chronic and recurrent pain periods, and their activities and quality of life are adversely affected. The causes of neck pain are not fully known. Long-term wrong static posture is considered as one of the most important causes of neck pain..

When studies examining the relationship between neck pain and spinal normality are investigated, it is seen that these studies mainly focus on the relationship between neck pain and cervical posture. In these studies, it is suggested that abnormal cervical lordosis and forward head posture are associated with neck pain development and its recurrence.

Although there are many studies examining the relationship between neck pain and the posture of the cervical region, studies investigating postural and angular changes in other parts of the spine in patients with neck pain are inadequate. In a review study, which stated that each segment of the spine is interrelated to other segments, it was mentioned that pelvis is associated with lumbar lordosis, lumbar lordosis is interrelated to thoracic kyphosis, and thoracic kyphosis has an impact on cervical lordosis. On the other hand, in this review study, it was emphasized that the relationship between pelvis and thoracic region decreases as the path from the pelvis to the cervical region becomes complicated. However, it is reported that when a postural disorder such as a decrease in lumbar lordosis and/or an increase in thoracic kyphosis occurs, the cervical lordosis increases as a compensatory mechanism.

Although it is known that the cervical, thoracic and lumbar regions of the spine are related with each other biomechanically, there are no studies examining the relationship between cervical pain and other regions of the spine. Lau et al. reported that the upper thoracic angle increases in patients with neck pain and this angle is a good predictor of neck pain.

Since the spine is a whole, it is thought that any deficiency at one end of the whole can affect other segments. Therefore, the purpose of this study was to examine angular changes of the spine and compare it with the control group according to the state of pain in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* presence of neck pain for at least 3 months
* absence of any other problems related to other parts of the spine such as low back pain
* absence of any neurological, rheumatical or musculoskeletal problems

Exclusion Criteria:

* history of spinal surgery
* inclusion in physiotherapy program in the last 6 months
* pregnancy
* risk of osteoporosis
* positive test of vertebrobasilar artery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who were referred to the physiotherapy program by a specialist physician (SS) and met the inclusion criteria were included in the study. Inclusion criteria were as follows: being 18-65 years old, presence of neck pain for at least 3 months, absence of any other problems related to other parts of the spine such as low back pain, absence of any neurological, rheumatical or musculoskeletal problems. Exclusion criteria were as follows: history of spinal surgery, inclusion in physiotherapy program in the last 6 months, pregnancy, risk of osteoporosis and positive test of vertebrobasilar artery. According to these criteria, 81 patients with chronic neck pain and 40 without any pain in their neck (as the control group) were included in the study. Individuals with neck pain were divided into 2 groups according to the severity of their pain. Individuals with neck pain score of 5 or less according to Visual Analogue Scale (VAS) were identified as Group 1, whereas those with any score
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2013-06-10 (Actual); Study Completion 2013-06-11 (Actual)

PRIMARY OUTCOMES:
Demographic data | baseline
  Demographic data (age, height, weight, body mass index (BMI) and duration of symptoms (duration of diagnosis)) of all individuals were recorded. All individuals were evaluated by the same researcher (OB) using the same test protocol.
Visual Analog Scale | baseline
  The severity of pain was evaluated by VAS. The average pain intensity in the last 4 weeks was questioned. The patients were asked to mark the severity of their pain on a 10-centimeter-long line where 0 stands for no pain and 10 for intolerable pain. The results were recorded in centimeter.
Thoracic and Lumbar Curvatures | baseline
  Thoracic and Lumbar Curvatures: Thoracic and lumbar region curvatures of individuals included in the study were evaluated by using Spinal Mouse (SM) (Idiag, Volkerswill, Switzerland). SM is a computer-aided electromechanical device that measures the curvatures of the spine at various postures. The locations marked on the skin were first determined by palpation and then marked with a cosmetic pen on the skin. The SM device was placed onto the 7th cervical vertebra and the recording started by pressing the button. Then the device was moved over the spinous processes of the spine from the 7th cervical vertebrae down to the 3rd sacral vertebrae where the button on the device was pressed again to finish the assessment. At a frequency of about 150 Hz, the device makes measurements along the spine at every 1.3 mm and records the data (The average length of the spine is 550 mm and the time required to measure the entire length is 2 to 4 seconds, so approximately 423 measurements are made in 3

CONTACTS AND LOCATIONS:
Overall Officials: ÖZNUR büyükturan, professor, Study Director — Kırşehir Ahi Evran Univercity

IPD SHARING:
Plan to Share IPD: Undecided